CLINICAL TRIAL: NCT02343874
Title: Impact of Alcohol Consumption of the General Population Who Visited Primary Health Care Centers on the Use of Health Care Resources in Catalonia.
Brief Title: Impact of Alcohol Consumption on Use of Health Care Resources
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut Catala de Salut (Other Government); Institut Català de la Salut (Other); Public Health Agency of Barcelona (Other); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Antoni Gual, Senior consultant, Hospital Clinic of Barcelona
Other Study IDs: 2013/8739
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Alcohol Consumption
Keywords: Alcohol consumption; Primary health care; health care costs; health service utilization
MeSH Terms: conditions — Alcohol Drinking; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alcohol consumption: Patients over 17 years old with alcohol consumption registered in the electronic medical record (31st December 2012).
  No intervention is going to be administered but exposure to alcohol will be analysed
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be done. The exposure of interest in this study is alcohol consumption in patients attended in primary health.

SUMMARY:
The prevalence of alcohol-related disorders in the general population is around 10%. The relationship between the use of healthcare services, costs and the amount of alcohol consumed by the general population is unknown. Because alcoholism is a major public health problem, it is significant to determine the prevalence of consumption of primary users and the relationship between the dose of alcohol and health care costs. This information may allow the implementation of preventive strategies to reduce consumption with the aim to reduce morbidity and healthcare expenditure.

A cross-sectional study will be carried out. Patients over 17 years old, treated at primary healthcare centers in Catalonia that have available data on alcohol consumption from January 2010 to December 2012 will be included. Clinical and sociodemographic data will be collected. Health service use and health care costs from 2013 will be collected from SIDIAP (The Information System for the Development of Research in Primary Care) database.

A positive relationship between grams of alcohol consumed per week and the use of resources and health expenditure will be expected and also the level of risk of alcohol consumption. There will be a descriptive analysis of the clinical data and sociodemographic variables. A multivariate analysis will be done to see the relationship between alcohol consumption and health care costs and health care service utilization.

DETAILED DESCRIPTION:
The aim of the study is to describe the association between alcohol consumption and the use of health care resources and the health care costs in Catalonia, which is a region of Spain.

A cross-sectional study was done. Patients recruited in the study were those attended in the primary health care whose alcohol consumption was registered in the electronic medical record between 1st of January 2011 to 31st of December 2012. At Baseline (31st of December 2012), sociodemographic data and clinical data was recorded, and health care utilization and costs were obtained from year 2013.

Two different registers were used for sociodemographic, clinical and health service utilization indicators and costs. Information on life style factors (alcohol and tobacco consumption, body mass index), demographic information like the ecologic MEDEA index, and sick-leave costs were obtained from the Information System for the Development of Research in Primary Care (SIDIAP) database. This clinical database has anonymized records of almost the 80% of the Catalan population. General practitioners can record alcohol consumption in two different ways (quantitative and categorical information). A quantitative variable defined as grams of alcohol per week and a categorical variable measuring the risk of alcohol consumption (none, low risk, risky drinker). The type of risk was defined as follows (No drinker; Low drinker (men who drinks <280g per week of alcohol or women who drinks <179g per week); Riky drinker (men who drinks >=280g per week or women who drinks >=170g per week of alcohol, or men who drinks more than 5 drinks per occasion, women who drinks more than 4 drinks per occasion; men who drinks <280g per week of alcohol or women who drinks <179g per week and at the same time work with heavy machinery or are taking medication that could interfere with alcohol)).

Sociodemographic data (age and sex and socioeconomic status) and clinical data (hypertension, diabetes, hyperlipemia, obesity, psychiatric diseases, clinical risk groups and diagnosis wholly attributable and partly attributable to alcohol) were obtained from the central register (Morbidity Register) provided by the Catalan Health service. From the same register data on health service utilization was collected. These indicators include: the number and costs of outpatients visits from doctor, nurse and social worker in primary health centres; hospital admissions, emergency room visits, mental health outpatients visits, and specialists referrals. Data on acute and chronic hospitalizations were analysed using three indicators: costs, number of admissions and hospital days, defined as the number of days stayed in any hospital. Three types of hospitals were included in the administrative system: general (acute) hospital, rehabilitation hospital and psychiatric hospital. The patient's diagnosis at admission was also registered. Using the same categories as Jones and colleagues, we distinguished between entry diagnosis wholly attributable to alcohol (e.g., alcohol dependence or alcoholic liver cirrhosis), entry diagnosis partly attributable (acute and chronic), or not related to alcohol. Also information about medication expenses and seak-leave costs were included.

Quality checks, in SIDIAP database, to identify duplicate patient identification are performed centrally at the time of each SIDIAP database update. Furthermore, checks for logic values are performed and unexpected values are dismissed. A part from that, a number of papers have been published on the validity of SIDIAP coding for various conditions. The quality and consistency of the central Catalan register is very good with a built-in validation to detect problems and inconsistencies between variables. In addition, the system is periodically externally validated to ensure quality of data, as these data are used to control payment to service providers.

Descriptive analyses of sociodemographic and clinical data will be carried out. Analysis of variance (ANOVA) and t-students tests will be used to compare continuous data, and chi-square analysis for categorical variables. Bonferroni correction will be used for multiple comparisons. A probability level of 5% or less will be considered as statistically significant. Poisson regression and sensitivity analyses with negative binomial regression will be done. Linear regression will be done to analyze the relationship between grams per week of alcohol and health costs. Data were analysed with Statistical Analysis Software.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 17 years old
* Patients with alcohol consumption registered in the medical record

Exclusion Criteria:

* patients <= 17 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 17 years old attended in the primary health care setting that have their alcohol consumption registered in the medical record.
Sampling Method: Non-Probability Sample
Enrollment: 1911771 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Health economic costs (composite measure) | 1 year
  Association between alcohol consumption and Health economic costs (euros per individual) which include the sum of the following costs: primary health costs (appointments with the doctor, nurse or social worker), laboratory costs, pharmacy expenses, Inpatients costs from General hospitals, Psychiatric hospitals or rehabilitation hospitals, costs due to emergency visits, costs of outpatient visits in mental health and costs due to appointments with specialists.
sick-leave costs | 1 year
  sick leave costs (euros per individual)

SECONDARY OUTCOMES:
Primary health care costs | 1 year
  Association between alcohol consumption and primary health care costs which include costs due to the patients appointments with the doctor, nurse or social worker (euros per individual)
laboratory costs | 1 year
  Association between alcohol consumption and laboratory costs (euros per individual)
Pharmacy expenses | 1 year
  Association between alcohol consumption and pharmacy expenses (euros per individual)
Inpatient costs | 1 year
  Association between alcohol consumption and inpatient costs which include: Inpatients costs from General hospitals, Psychiatric hospitals or rehabilitation hospitals (euros per individual)
costs due to emergency attendance | 1 year
  Association between alcohol consumption and costs due to the emergency room attendance (euros per individual)
outpatient mental health costs | 1 year
  Association between alcohol consumption and outpatients mental health costs (euros per individual).
specialists consults costs | 1 year
  Association between alcohol consumption and costs due to specialists consults
Primary health visits | 1 year
  Association between alcohol consumption and the number of appointments with the general practitioner, nurse or social worker
Admissions in hospital | 1 year
  Association between alcohol consumption and the number of hospital admissions (general hospital, mental health and rehabilitation hospitals)
days of stay in hospital | 1year
  Association between alcohol consumption and the number of days of stay in hospitals (General Hospital, Psychiatric Hospital or Rehabilitation hospital)
emergency contacts | 1 year
  Association between alcohol consumption and the number of emergency visits.
specialists appointments | 1 year
  Association between alcohol consumption and the number of visits done with a specialist.
Hospital admissions causes | 1 year
  Number of hospital admissions depending on the cause (wholly attributable to alcohol, partly attributable- acute, partly attributed-chronic or not related with alcohol consumption)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gual, PhD, Principal Investigator — Institut d'investigacions Biomèdiques Agust Pi i Sunyer (IDIBAPS)
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Anderson P, Cremona A, Paton A, Turner C, Wallace P. The risk of alcohol. Addiction. 1993 Nov;88(11):1493-508. doi: 10.1111/j.1360-0443.1993.tb03135.x. PMID 8286995
- [Background] Compton WM, Thomas YF, Stinson FS, Grant BF. Prevalence, correlates, disability, and comorbidity of DSM-IV drug abuse and dependence in the United States: results from the national epidemiologic survey on alcohol and related conditions. Arch Gen Psychiatry. 2007 May;64(5):566-76. doi: 10.1001/archpsyc.64.5.566. PMID 17485608
- [Background] Laramee P, Kusel J, Leonard S, Aubin HJ, Francois C, Daeppen JB. The economic burden of alcohol dependence in Europe. Alcohol Alcohol. 2013 May-Jun;48(3):259-69. doi: 10.1093/alcalc/agt004. Epub 2013 Jan 30. PMID 23371284
- [Background] Rehm J, Giesbrecht N, Patra J, Roerecke M. Estimating chronic disease deaths and hospitalizations due to alcohol use in Canada in 2002: implications for policy and prevention strategies. Prev Chronic Dis. 2006 Oct;3(4):A121. Epub 2006 Sep 15. PMID 16978496
- [Background] Gual A, Lligona A, Costa S, Segura L, Colom J. [Long term impact of treatment in alcoholics. Results from a 10-year longitudinal follow-up study of 850 patients]. Med Clin (Barc). 2004 Sep 25;123(10):364-9. doi: 10.1016/s0025-7753(04)74520-0. Spanish. PMID 15482699
- [Background] Gual A, Bravo F, Lligona A, Colom J. Treatment for alcohol dependence in Catalonia: health outcomes and stability of drinking patterns over 20 years in 850 patients. Alcohol Alcohol. 2009 Jul-Aug;44(4):409-15. doi: 10.1093/alcalc/agp032. Epub 2009 Jun 2. PMID 19491281
- [Background] Geary T, O'Brien P, Ramsay S, Cook B; Scottish Intensive Care Trainees' Audit Share Group. A national service evaluation of the impact of alcohol on admissions to Scottish intensive care units. Anaesthesia. 2012 Oct;67(10):1132-7. doi: 10.1111/j.1365-2044.2012.07233.x. Epub 2012 Jul 16. PMID 22804562
- [Background] Lawder R, Grant I, Storey C, Walsh D, Whyte B, Hanlon P. Epidemiology of hospitalization due to alcohol-related harm: evidence from a Scottish cohort study. Public Health. 2011 Aug;125(8):533-9. doi: 10.1016/j.puhe.2011.05.007. Epub 2011 Jul 26. PMID 21794884
- [Background] Taylor B, Rehm J, Patra J, Popova S, Baliunas D. Alcohol-attributable morbidity and resulting health care costs in Canada in 2002: recommendations for policy and prevention. J Stud Alcohol Drugs. 2007 Jan;68(1):36-47. doi: 10.15288/jsad.2007.68.36. PMID 17149516
- [Background] McKenny M, O'Beirne S, Fagan C, O'Connell M. Alcohol-related admissions to an intensive care unit in Dublin. Ir J Med Sci. 2010 Sep;179(3):405-8. doi: 10.1007/s11845-010-0498-y. Epub 2010 May 28. PMID 20509003
- [Background] Corrao G, Bagnardi V, Zambon A, Arico S. Exploring the dose-response relationship between alcohol consumption and the risk of several alcohol-related conditions: a meta-analysis. Addiction. 1999 Oct;94(10):1551-73. doi: 10.1046/j.1360-0443.1999.9410155111.x. PMID 10790907
- [Background] Hvidtfeldt UA, Rasmussen S, Gronbaek M, Becker U, Tolstrup JS. Influence of smoking and alcohol consumption on admissions and duration of hospitalization. Eur J Public Health. 2010 Aug;20(4):376-82. doi: 10.1093/eurpub/ckp153. Epub 2009 Sep 30. PMID 19793836
- [Background] Cohen E, Feinn R, Arias A, Kranzler HR. Alcohol treatment utilization: findings from the National Epidemiologic Survey on Alcohol and Related Conditions. Drug Alcohol Depend. 2007 Jan 12;86(2-3):214-21. doi: 10.1016/j.drugalcdep.2006.06.008. Epub 2006 Aug 17. PMID 16919401
- [Background] Baser O, Chalk M, Rawson R, Gastfriend DR. Alcohol dependence treatments: comprehensive healthcare costs, utilization outcomes, and pharmacotherapy persistence. Am J Manag Care. 2011 Jun;17 Suppl 8:S222-34. PMID 21761948
- [Background] Bray JW, Cowell AJ, Hinde JM. A systematic review and meta-analysis of health care utilization outcomes in alcohol screening and brief intervention trials. Med Care. 2011 Mar;49(3):287-94. doi: 10.1097/MLR.0b013e318203624f. PMID 21263359
- [Background] Kaner EF, Dickinson HO, Beyer F, Pienaar E, Schlesinger C, Campbell F, Saunders JB, Burnand B, Heather N. The effectiveness of brief alcohol interventions in primary care settings: a systematic review. Drug Alcohol Rev. 2009 May;28(3):301-23. doi: 10.1111/j.1465-3362.2009.00071.x. PMID 19489992
- [Background] Kaner EF, Beyer F, Dickinson HO, Pienaar E, Campbell F, Schlesinger C, Heather N, Saunders J, Burnand B. Effectiveness of brief alcohol interventions in primary care populations. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004148. doi: 10.1002/14651858.CD004148.pub3. PMID 17443541
- [Background] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Background] Garcia-Gil Mdel M, Hermosilla E, Prieto-Alhambra D, Fina F, Rosell M, Ramos R, Rodriguez J, Williams T, Van Staa T, Bolibar B. Construction and validation of a scoring system for the selection of high-quality data in a Spanish population primary care database (SIDIAP). Inform Prim Care. 2011;19(3):135-45. doi: 10.14236/jhi.v19i3.806. PMID 22688222